CLINICAL TRIAL: NCT06991998
Title: Evaluation of Clinical and Radiological Outcomes Following the Treatment of Periodontal Intraosseous Defects Using Autogenous Tooth-derived Graft or Autogenous Bone Graft With Enamel Matrix Derivatives. A 12-month Randomized Controlled Clinical Trial.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Forgó Kristóf, Periodontist, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200/2024.
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis
Keywords: periodontal regeneration; periodontitis; graft; intrabony defect; tooth-derived graft; enamel matrix derivatives; autogenous bone graft
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autogenous Bone Graft + EMD (Active Comparator)
  Interventions: Procedure: Autogenous bone graft with enamel matrix derivative
- Autogenous Tooth-Derived Graft + EMD (Experimental)
  Interventions: Procedure: Autogenous tooth-derived graft with enamel matrix derivative

INTERVENTIONS:
Procedure: Autogenous bone graft with enamel matrix derivative — Participants receive periodontal regenerative surgery using autogenous bone graft harvested from a secondary intraoral donor site (mandibular ramus or maxillary tuberosity) with a bone scraper. The bone graft is placed into the debrided intraosseous defect, and enamel matrix derivative (EMD) is applied to the root surface. Surgical access is performed using a single flap approach (SFA), and primary closure is achieved with microsurgical sutures.
  Arms: Autogenous Bone Graft + EMD
Procedure: Autogenous tooth-derived graft with enamel matrix derivative — Participants receive periodontal regenerative surgery using autogenous tooth-derived particulate graft processed from an extracted tooth using a standardized protocol (Bonmaker® device and chemical decontamination), combined with enamel matrix derivative (EMD) applied to the root surface. The surgical site is accessed using a single flap approach (SFA), and graft material is placed into the non-self-contained intraosseous defect after debridement. Primary closure is achieved with microsurgical sutures.
  Arms: Autogenous Tooth-Derived Graft + EMD

SUMMARY:
This clinical study aims to evaluate and compare two different materials used to treat bone defects caused by periodontitis. Periodontitis is a chronic inflammatory condition that damages the supporting structures of teeth, including the bone. One of the most severe forms of this damage is called an "intraosseous defect," where the bone around a tooth is lost in a vertical pattern.

To repair these defects, dentists often perform a regenerative surgery using grafting materials and biologically active substances to stimulate tissue regrowth. The current standard includes using autogenous bone grafts (ABG)-bone taken from another part of the patient's mouth-combined with enamel matrix derivatives (EMD), a protein-based gel that promotes healing. However, this approach requires creating a second surgical site to harvest the bone, which can increase patient discomfort and healing time.

Recently, a promising alternative has emerged: autogenous tooth-derived bone grafts (ATB). In this technique, a patient's own extracted tooth is processed into a grafting material and used to fill the bone defect. This method has the advantage of using a material that would otherwise be discarded and avoids the need for an additional surgical area. Early studies suggest that tooth-derived grafts may have similar regenerative potential to traditional bone grafts because of their comparable structure and the presence of natural growth factors.

The purpose of this randomized controlled trial is to determine whether ATB combined with EMD can achieve the same or better clinical and radiological outcomes as ABG combined with EMD in the treatment of periodontal intraosseous defects.

A total of 60 adult patients with chronic periodontitis will be enrolled. Each participant must have at least one advanced bone defect around a tooth and one other tooth that needs to be extracted for unrelated reasons. Patients will be randomly assigned to receive either ATB or ABG, both with EMD, during a single surgical procedure.

The study includes multiple follow-up visits over the course of one year, and at 12 months, a re-entry surgery will allow the research team to directly observe bone healing inside the defect.

The findings could support a more patient-friendly and equally effective alternative to traditional bone grafting in periodontal regenerative surgery.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the regenerative efficacy of autogenous tooth-derived graft material (ATB) in comparison with autogenous bone graft (ABG) in the treatment of periodontal intraosseous defects. Enamel matrix derivative (EMD) is applied to all defects in both treatment groups as part of the regenerative procedure, and a standardized, minimally invasive flap approach is used for defect access.

The regenerative management of intrabony periodontal defects often involves the application of biologically active materials in conjunction with particulate grafts, especially in non-contained defects. While autogenous bone is widely regarded as the gold standard due to its osteogenic and osteoinductive properties, its harvesting requires an additional surgical site, leading to increased morbidity and treatment time. Autogenous tooth-derived biomaterial (ATB) represents an innovative alternative with promising biological properties. The dentin graft contains a variety of growth factors and has demonstrated regenerative potential in preclinical and clinical studies.

In this study, eligible defects are treated surgically using the Single Flap Approach (SFA), either buccally or palatally/lingually, depending on defect location. After local anesthesia, a full-thickness mucoperiosteal flap is elevated using sulcular incisions extended to adjacent teeth, while preserving the interdental papilla. The defect area is thoroughly debrided and root surfaces are conditioned with 24% EDTA gel (PrefGel®, Straumann) for 2 minutes, followed by thorough rinsing with sterile saline. Then, enamel matrix derivative (Emdogain®, Straumann) is applied onto the root surface according to the manufacturer's instructions.

In the test group, autogenous tooth-derived graft is prepared using the Bonmaker® system (Korean Dental Solution). The patient's extracted tooth is cleaned and processed into particulate form. A decalcification and sterilization process is carried out in a closed system, ensuring the preservation of bioactive molecules including TGF-β, BMPs, and IGFs. In the control group, autogenous bone is harvested from intraoral donor sites such as the mandibular ramus or maxillary tuberosity using a manual bone scraper. The graft material is applied into the defect without the use of a barrier membrane.

Flaps are repositioned and sutured using 6-0 monofilament non-resorbable sutures, employing horizontal mattress and interrupted techniques to ensure tension-free primary closure. Postoperative care includes systemic antibiotics (amoxicillin/clavulanic acid or clindamycin in case of allergy) for 7 days, analgesics as needed, and 0.2% chlorhexidine mouthrinse twice daily for 14 days. Sutures are removed after 10 to 14 days. Supportive periodontal therapy is provided monthly for the first 3 months, then every 2 to 3 months until the final follow-up.

Radiographic evaluation is standardized using the long cone paralleling technique and individualized silicone bite registrations. Radiographs are obtained preoperatively and at 6 and 12 months following the surgical intervention.

A re-entry procedure is performed 12 months postoperatively to allow for direct clinical evaluation of bone fill. Custom-made acrylic templates are fabricated to standardize probing during the initial surgery and the re-entry.

The objective of the study is to determine whether autogenous tooth-derived biomaterial can achieve comparable regenerative outcomes to autogenous bone graft, while offering the advantage of reduced patient morbidity and surgical complexity.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic periodontitis
* Both male and female participants
* Patients with less than 25% plaque score (FMPS: Full Mouth Plaque Score) and bleeding index (FMBS: Full Mouth Bleeding Score) after non-surgical periodontal therapy
* Good patient compliance (maintains good oral hygiene and is willing to participate in 12-month follow-up)
* Patients who understand the nature of the study after receiving written information and provide signed informed consent
* Patients older than 18 years
* Non-self-contained intraosseous defects (wide (radiological angle > 37°) and/or one- or two-wall defects) in the maxilla or mandible with a baseline probing depth of ≥ 6 mm
* The defect has an intraosseous component of ≥ 3 mm
* The patient has at least one tooth that needs extraction for any reason

Exclusion Criteria:

* Patients with systemic conditions such as:

Alcoholism Drug addiction Known HIV, HBV, or HCV infection Patients undergoing chemotherapy or radiation therapy Current or past head and neck radiation therapy Untreated insulin-dependent diabetes mellitus Clinically significant osteoporosis or other systemic conditions affecting bone metabolism Clinically significant cardiovascular conditions such as decompensated heart failure, hemodynamically significant heart valve insufficiency, or myocardial infarction within the last 3 months Clinically significant coagulation disorders

* Previous or current systemic corticosteroid therapy (within 2 months of inclusion): more than 5 mg of prednisolone per day
* Previous or current bisphosphonate therapy lasting at least 30 days within the past 12 months
* Long-term antibiotic or anti-inflammatory therapy within the past 4 months
* Pregnant or breastfeeding women
* Smoking (>5 cigarettes/day)
* Furcation involvement
* Wisdom teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-10-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | At baseline and at 6 months and 12 months following the surgical intervention

SECONDARY OUTCOMES:
Bone fill in the intraosseous defects | During the surgical intervention and after 12 months during the re-entry
Postoperative pain level | 7 days from the surgical intervention
  Using Visual Analog Scale (VAS)
Clinical attachment gain (∆CAL) | At baseline and at 6 months and 12 months following the surgical intervention
Changes in gingival recession (∆GR) | At baseline and at 6 months and 12 months following the surgical intervention
Radiological bone fill | At baseline and at 6 months and 12 months following the surgical intervention
  Standardized intraoral radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Department of Periodontology, Budapest, Budapest, Hungary